CLINICAL TRIAL: NCT04390815
Title: Effect of Insulin on Wound Healing- A Randomized Controlled Trial
Brief Title: Effect of Insulin on Wound Healing-A Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Bahrain (Other Government)
Responsible Party: Principal Investigator, Abeer AlSaweer, Central Diabetes clinic coordinator in PHC, Ministry of Health, Bahrain
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IWCT20
Record Dates: First submitted 2020-04-26; First posted 2020-05-18 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Wound Heal
MeSH Terms: interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Before starting the therapeutic procedure, all wounds will be fully washed with normal saline.
  Group A patients will receive 10 units (0.1 mL) of regular insulin (manufactured by novo nordisk) in solution with 1 cc of normal saline 0.9% for each 10 cm of wound. The solution will be sprayed on the wound surface with an insulin syringe needle, once daily.
  The patients in this arm will receive conventional therapy.
  Interventions: Drug: Insulin
- Control (Placebo Comparator): Before starting the therapeutic procedure, all wounds will be fully washed with normal saline Group B patients will receive conventional topical application without insulin
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Adding insulin to conventional wound treatment
  Other Names: Regular Insulin

SUMMARY:
A randomized controlled trial examining the effect of insulin on wound healing in both diabetics and non diabetic patients in a local health center in Bahrain.

DETAILED DESCRIPTION:
This is a double blinded RCT comparing the effect of insulin on wound healing in both diabetics and non diabetics.

The study will run in primary care setting in Bahrain. The aim of this study is to heal wound in an innovative way. and the Objective: to evaluate the effect of topical insulin administration on wound healing.

All adult patients with skin wounds attending primary health care center will be included in the study. Patients with acute and chronic wounds of the upper and lower extremities will be eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Texas 1 and 2 wound criteria

Exclusion Criteria: Texas 3 and 4 wound criteria

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Area of wound healing | 4 months
  Rate of wound healing will be calculated as the difference between the primary and final wound area in mm as a function of healing time (in days) and reported as mm/day.

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 4 months

REFERENCES:
- [Derived] Xue Y, Reddy SK, Garza LA. Toward Understanding Wound Immunology for High-Fidelity Skin Regeneration. Cold Spring Harb Perspect Biol. 2022 Jul 1;14(7):a041241. doi: 10.1101/cshperspect.a041241. PMID 35667792